CLINICAL TRIAL: NCT06522399
Title: Outcome of Transanal Minimally Invasive (TAMIS) Mucosal Resection in Patients With Obstructed Defecation Syndrome - a Pilot Study
Brief Title: Outcome of TAMIS Mucosal Resection in Patients With ODS
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Dr. Christopher Dawoud, Medical University of Vienna
Other Study IDs: 1415/2022
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Constipation, Impaction, and Bowel Obstruction; TAMIS Mucosectomy; Obstructed Defecation Syndrome
Keywords: obstructed defecation syndrome; TAMIS mucosectomy
MeSH Terms: conditions — Constipation; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with obstructed defecation who undergo TAMIS mucosectomy: patients with obstructed defecation and rectocele or intussuception
  Interventions: Procedure: TAMIS mucosectomy

INTERVENTIONS:
Procedure: TAMIS mucosectomy — internal Delorme's procedure using TAMIS

SUMMARY:
Patients, aged 18 - 90 years, undergoing TAMIS mucosectomy at the Department of General Surgery at the Medical University of Vienna are enrolled into our study.

Primary endpoint is the outcome (improvement of ODS symptoms), defined by ODS score.

DETAILED DESCRIPTION:
Various surgical approaches for the treatment of obstructed defecation syndrome (ODS) commonly associated with rectocele and rectal intussusception have been investigated in the literature. Methods such as stapled transanal resection of the rectum (STARR) and ventral prosthesis rectopexy (VPR) show promising results at least in the short term. In the long-term, however, the results do not seem convincing. Schiano di Visconte et al. report a recurrence of ODS symptoms in 40 percent of the patients, treated with stapled transanal rectal resection in a 10-year follow up. The clinical outcome of surgical treatment of ODS using transanal minimally invasive surgery (TAMIS) in the sense of a mucosal resection without stapling technique has not yet been investigated. This project is designed to show the short-term outcome of non-stapled mucosal resection through TAMIS.

ELIGIBILITY:
Inclusion Criteria:

* Need of minimal invasive mucosal resection due to obstructed defecation syndrome after several unsuccessful conservative treatments over a period of more than 6 months with presence of an organic cause (Symptomatic intussusception with or without rectocele) in medical examinations (defecography, endoluminal ultrasound, endoanal manometry)
* Age: 18-90 years
* Ability and willingness to understand and comply with planned interventions during the study.
* Voluntarily signed informed consent after a full explanation of the study to the participant.

Exclusion Criteria:

* Any physical or mental disorder could interfere with the participant's safety during the clinical trial or with the study objectives.
* Inability to communicate well with the investigator due to language problems or reduced mental development.
* Inability or unwillingness to give written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled who ungergo minimally invasive mucosal resection due to obstructed defecation syndrome after several unsuccessful conservative treatments over a period of more than 6 months with presence of an organic cause (Symptomatic intussusception with or without rectocele) in medical examinations (defecography, endoluminal ultrasound, endoanal manometry)
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
functional outcome assessment | 6 months
  functional outcome defined by ODS score

SECONDARY OUTCOMES:
fecal incontinence assessment | 6 months
  fecal incontinence improvement or worsening measured by using the VAIZEY Score
Quality of life assessment | 6 months
  Health-related quality of life after TAMIS in ODS patients, defined by Quality of Life Score (SF12).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, MD, Study Chair — Medical University of Vienna, Head of Pelvic Floor surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD can be shared just in anonymised form in case of an ethical agreement with other researchers.